CLINICAL TRIAL: NCT06392971
Title: A Randomized Control Study of Deep-sea Fish Oil for Prevention of Acute Radiation-induced Esophagitis in Patients With Esophageal Cancer
Brief Title: Deep-sea Fish Oil for Prevention of Acute Radiation-induced Esophagitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23LCYJ049
Record Dates: First submitted 2024-04-25; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Radiation Toxicity; Esophagitis; Esophageal Cancer
Keywords: Fish oil; Acute Radiation-induced Esophagitis; Esophageal Cancer; prevention
MeSH Terms: conditions — Radiation Injuries; Esophagitis; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, randomized controlled clinical study. The present study intends to continuously enroll 120 patients with esophageal cancer who are to receive radiotherapy, and randomly divide the enrolled patients into two groups. One group receive treatment of deep-sea fish oil and the other group is blank control. The differences of ARIE occurrence, ARIE degree, pain degree, and the changes of the inflammatory index were compared.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preventive use of deep-sea fish oil (Experimental)
  Interventions: Drug: Deep-sea fish oil
- Preventive use of placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Deep-sea fish oil — Starting from radiotherapy, the whole course of prophylactic oral deep-sea fish oil should be taken at the recommended dosage of 1g po bid according to the instructions (the administration method is to take it with the drug, remove the film on the drug surface, slowly swallow it in a supine position, and make the liquid fully contact with the esophageal mucosa). If no acute radioactive esophagus was assessed during the course of treatment, the patient was administered orally until the end of radiotherapy. If the patient developed radioactive esophagitis during the course of treatment, the relevant outcome measures were recorded and used as the endpoint event of the phase I study. The end point for patients without acute radiation esophagitis was at the completion of radiation therapy.
  Arms: Preventive use of deep-sea fish oil
Other: Placebo — Take a capsule made of food oil that looks like deep-sea fish oil at a dose of 1g po bid. Treatment is discontinued when patients develop acute radiation esophagitis.
  Arms: Preventive use of placebo

SUMMARY:
Purpose：To observe and evaluate the clinical efficacy and safety of deep-sea fish oil in preventing acute radiation-induced esophagitis (ARIE).

Methods and Materials：A total of 120 patients with esophageal cancer treated with radiotherapy were randomly assigned (1:1) to treatment or control group. In the treatment group, 1g deep-sea fish oil was oral administrated prophylactically twice a day，the control group was blank control. The clinical efficacy of deep-sea fish oil on prevention of ARIE was evaluated by comparing the differences in the occurrence time, the grade and incidence of ARIE. Additionally, the change in nutritional status was also investigated. Hemanalysis, liver function, kidney function changes， and adverse reactions were compared before and after treatment to evaluate the safety of deep-sea fish oil.

DETAILED DESCRIPTION:
Radiotherapy is an important treatment for esophageal cancer, and acute radiation-induced esophagitis (ARIE) is the most common complication during radiotherapy. The present study was conducted to investigate the clinical efficacy of deep-sea fish oil in the prevention and treatment of ARIE, and to evaluate the effects of deep-sea fish oil on patients' nutritional status, quality of life, pain management, and the effect on the treatment. This is a prospective, single-center, randomized controlled clinical study. The present study has been registered in the Chinese Clinical Trials Registry (ChiCTR2200056847). The present study intends to continuously enroll 120 patients with esophageal cancer who are to receive radiotherapy, and randomly divide the enrolled patients into two groups. One group receive treatment of deep-sea fish oil and the other group is blank control. The differences of ARIE occurrence, ARIE degree, pain degree, and the changes of the inflammatory index were compared.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, ≤70 years old, gender is not limited;
2. Histological or cytological evidence of esophageal, lung, or breast cancer;
3. ECOG score of 0-2, no swallowing pain or severe dysphagia before radiotherapy;
4. Liver and kidney function, bone marrow function and cardiopulmonary function are not contraindicated by radiotherapy and chemotherapy;
5. PG-SGA score <9;
6. Not pregnant or breastfeeding;
7. The subject must understand and sign the informed consent
8. Have reading comprehension ability and can complete the questionnaire with medical assistance;
9. Those who voluntarily participate in the study and sign the informed consent letter in person.

Exclusion Criteria:

1. Prior radiation therapy;
2. Patients with severe underlying diseases, who cannot tolerate radiotherapy and chemotherapy due to severe liver and kidney insufficiency and poor cardiopulmonary function;
3. Pregnant or lactating female patients;
4. Suffering from severe mental illness and poor compliance;
5. Other cases deemed unsuitable for inclusion by the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
The duration from initiation of radiotherapy to the onset of acute radiation esophagitis | Approximately 2 months
Severity of acute radiation esophagitis | Approximately 2 months
  Using the Radiation Therapy Oncology Group (RTOG) grading method for radiation esophagitis, patients with acute radiation esophagitis are evaluated daily from the first day onwards. Specifically, level 0: asymptomatic; Grade I: mild dysphagia or pain in swallowing, requiring topical or non-narcotic analgesia; Grade II: moderate dysphagia or swallowing pain, requiring narcotic analgesia; Grade III: severe dysphagia or dysphagia pain, accompanied by dehydration or weight loss greater than 15%, requiring a nasal feeding diet with intravenous fluids or high nutrients; Grade IV: complete obstruction, accompanied by ulceration, perforation, and fistula.
Incidence of severe acute radiation esophagitis | Approximately 2 months

SECONDARY OUTCOMES:
Pain degree | Approximately 2 months
  For patients with acute radiation esophagitis in the two groups, the Numerical Rating Scale (NRS) pain scoring method was used to evaluate the pain degree daily from the first day of acute radiation esophagitis, which was usually divided into the following criteria: 0 score: no pain 2; Scores 1-3: mild pain; 4-6 points: moderate pain; Score 7-10: Severe pain. The NRS score is based on a 10-point scale of pain, and the patient makes a numerical score to let the doctor know the level and level of pain.
The concentration of plasma C-reactive protein | Approximately 2 months
  The concentrations of plasma C-reactive protein were measured at three-time points at the beginning of radiotherapy, completion of 10 fractionated radiotherapy, and completion of 20 fractionated radiotherapy.
The concentration of plasma IL-6 | Approximately 2 months
  The concentrations of plasma IL-6 were measured at the beginning of radiotherapy, completion of 10 fractionated radiotherapy, and completion of 20 fractionated radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chengdu Medical College, Chengdu, China

IPD SHARING:
Plan to Share IPD: No